CLINICAL TRIAL: NCT02247505
Title: A Randomized, Open-label, Multiple Dosing, 2-way Crossover Study to Evaluate the Pharmacokinetic Effect of Tadalafil on Tamsulosin in Healthy Male Volunteers
Brief Title: CKD-397 Drug-drug Interaction Study (B)
Acronym: CKD-397DDI(B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 150DDI14013
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Healty Male Volunteers
MeSH Terms: interventions — Tamsulosin; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1: Treatment A + Treatment B, PO (Other): Treatment A : Tamsulosin 0.2mg*1t for 5days, Treatment B : Tamsulosin 0.2mg*1t/day and Tadalafil 5mg*1t/day for 5days, Each treatment period was separated by a washout period of at least 10 days.
  Interventions: Drug: Harnal-D Cap. 0.2mg; Drug: Cialis Tab. 5mg
- Group2: Treatment B + Treatment A, PO (Other): Treatment A : Tamsulosin 0.2mg*1t for 5days, Treatment B : Tamsulosin 0.2mg*1t/day and Tadalafil 5mg*1t/day for 5days, Each treatment period was separated by a washout period of at least 10 days.
  Interventions: Drug: Harnal-D Cap. 0.2mg; Drug: Cialis Tab. 5mg

INTERVENTIONS:
Drug: Harnal-D Cap. 0.2mg
  Other Names: Tamsulosin 0.2mg
Drug: Cialis Tab. 5mg
  Other Names: Tadalafil 5mg

SUMMARY:
The purpose of this study is to investigate to effect of tadalafil on the pharmacokinetic properies of tamsulosin

DETAILED DESCRIPTION:
This study is a randomized, open-label, mutiple dosing, 2-way crossover design to evaluate the pharmacokinetic effect of tadalafil(5mg) on tamsulosin(0.2mg) in healthy male subjects Subjects will receive repeated dose of tamsulosin (0.2mg*1t/day) or tamsulosin (0.2mg*1t/day) / tadalafil (5mg*1t/day) for 5days Each treatment period was separated by a washout period of at least 10 days. Each period of study will enroll 14 healthy male subjects. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate, safety laboratory data, and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man age 19 years or more and less than 55 years old at the time of screening.
* BMI more than 17.5kg / m2 and less than 30.5kg / m2 and weight more than 55kg
* Subject without congenital or chronic diseases and no psychotic symptoms or findings from the medical examination.
* Suitable subject who is determined by laboratory tests such as hematology tests, blood chemistry, urinalysis test according to the characteristics of the drug and screening tests such as ECG test.
* Subject who fully understand the clinical trials after in-depth explanation given prior to the clinical study, decided to join the clinical trials by their will and signed consent form which approved by Chonbuk National University Hospital IRB.
* Subjects who are able to comply with all scheduled visits, laboratory tests and other procedures.

Exclusion Criteria:

* Subject who has a history of blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic diseases that is clinically significant (Except untreated asymptomatic seasonal allergies at the time of administration)
* Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption.
* Showing the value that corresponds to following laboratory parameters: AST or AST > 2* upper limit of normal range.
* Alcohol > 210g/week, within 6 months prior to the screening.
* Taking the medication involved in other clinical trials within two months before the first dose medication characters.
* Sitting Systolic Blood Pressure ≥ 140 mmHg, Diastolic Blood Pressure ≥ 90 mmHg at the time of screening.
* History of alcohol or drug abuse, within 1 year
* Positive result in urine drug test(Amphetamines, Cocaine, Opioid, Benzodiazepines, Cannabinoid)
* Positive result in Serology test(Hepatitis B, Hepatitis C, HIV(Human Immunodeficiency Virus), TPPA(qual)).
* Subject who takes an abnormal meal which can affect the ADME of drug.
* Subjects who treated with metabolizing enzyme inducers or inhibitors such as barbitals within 30days prior to the first dosing.
* Smoker (> 20cigarettes/day)
* Subjects who takes ETC or OTC medicine within 10days before the first IP administration.
* Subject who done the whole blood donation within two months or component blood donation within 1 month prior to the first dosing.
* Subject who can increase risk due to clinical test and administration of drugs or has Severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
* Subject with taking any forms of organic nitrate periodically and/or intermittently.
* Subject with known hereditary degenerative retinal disease including retinitis pigmentosa.
* Subject with serious history of hypersensitivity or allergy to investigational product.
* Subject who Lost sight of one eye by Non-arteritic anterior ischemic optic neuropathy (NAION).
* Subject with genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption.
* Orthostatic hypotension
* Subjects who is not able to comply with guidelines described in the protocol.
* Subjects who is determined by investigator's decision as unsuitable for clinical trial participation.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tamsulosin AUCt(0-24) | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin Cmax | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h

SECONDARY OUTCOMES:
Tamsulosin Css,min | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin Css,av | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin Tss,max | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin t1/2 | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin CL/F | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin Vd/F | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin fluctuation[(Css,max-Css,min)/Css,av] | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h
Tamsulosin swing[(Css,max-Css,min)/Css,min] | 1D 0h, 3D 0h, 4D 0h, 5D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul Kim, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea